CLINICAL TRIAL: NCT02749162
Title: Perineural Dexamethasone Administered in Femural Nerve Block After Anterior Cruciate Ligament Reconstruction
Brief Title: Perineural Dexamethasone in Femural Nerve Block After Ligament Reconstruction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Foisor Orthopedics Clinical Hospital (Other)
Responsible Party: Principal Investigator, Munteanu Ana Maria, MD, PhD, MD PhD, Foisor Orthopedics Clinical Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ID AN-001-14
Record Dates: First submitted 2016-02-22; First posted 2016-04-22 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-08

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — dexamethasone 21-phosphate; Calcium Dobesilate; Acetaminophen; Morphine; Lidocaine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Placebo Comparator): After the spinal anesthesia regressed, the investigators performed a single shot femoral block with ropivacaine 0,5% 200 mg + lidocaine 1% 200 mg. After the block regression, at the first analgetic request the patients received the analgesia protocol was started for 24 h with paracetamol 1 g IV every 8 h and lornoxicam 8 mg PO every 12 h; if VAS was still over 3 after 30 min, morphine was given as a loading bolus of 0.1 mg/kg IV supplemented with 2 mg IV every 5 minutes until VAS <3. After 2 h morphine was administered SC ½ of the total loading dose at request.
  Interventions: Drug: Paracetamol; Drug: Morphine; Drug: Lidocaine; Drug: Ropivacaine
- Group B (Active Comparator): After the spinal anesthesia regressed, the investigators performed a single shot femural block with ropivacaine 0,5% 200 mg + lidocaine 1% 200 mg and 4 mg dexamethasone phosphate. After the block regression, at the first analgetic request the patients received the analgesia protocol was started for 24 h with paracetamol 1 g IV every 8 h and lornoxicam 8 mg PO every 12 h; if VAS was still over 3 after 30 min, morphine was given as a loading bolus of 0.1 mg/kg IV supplemented with 2 mg IV every 5 minutes until VAS <3. After 2 h morphine was administered SC ½ of the total loading dose at request.
  Interventions: Drug: Dexamethasone phosphate; Drug: Paracetamol; Drug: Morphine; Drug: Lidocaine; Drug: Ropivacaine
- Group C (Active Comparator): After the spinal anesthesia regressed, the investigators performed a single shot femural block with ropivacaine 0,5% 200 mg+ lidocaine 1% 200 mg and 8 mg dexamethasone phosphate.After the block regression, at the first analgetic request the patients received the analgesia protocol was started for 24 h with paracetamol 1 g IV every 8 h and lornoxicam 8 mg PO every 12 h; if VAS was still over 3 after 30 min, morphine was given as a loading bolus of 0.1 mg/kg IV supplemented with 2 mg IV every 5 minutes until VAS <3. After 2 h morphine was administered SC ½ of the total loading dose at request.
  Interventions: Drug: Dexamethasone phosphate; Drug: Paracetamol; Drug: Morphine; Drug: Lidocaine; Drug: Ropivacaine

INTERVENTIONS:
Drug: Dexamethasone phosphate — At the end of surgery the patients received single shot VIB block with the mixture according to the group allocation
  Other Names: Decadron
  Arms: Group B; Group C
Drug: Paracetamol — After the block regression, at the first analgetic request the patients received the analgesia protocol
  Other Names: Perfalgan
Drug: Morphine — After the block regression, at the first analgetic request the patients received the analgesia protocol
  Other Names: Morphine Sulfate
Drug: Lidocaine — At the end of surgery the patients received single shot VIB block with the mixture according to the group allocation
  Other Names: Xylocaine
Drug: Ropivacaine — At the end of surgery the patients received single shot VIB block with the mixture according to the group allocation
  Other Names: Naropin

SUMMARY:
The effect of perineural dexamethasone administered as an adjuvant in prolonging the duration of analgesia continues to be under debate. The investigators performed a prospective randomized study to evaluate the effect of perineural dexamethasone in different concentrations in postoperative analgesia in femoral nerve block for anterior cruciate ligament reconstruction.

DETAILED DESCRIPTION:
After Ethics committee approval, 75 patients American Society of Anesthesiologists score (ASA) I-III were randomized at the end of surgery into 3 groups of 25 patients each who underwent femoral nerve block: group A with 20 ml ropivacaine 0,5% and 20 ml lidocaine 1%; group B with 20 ml ropivacaine 0,5%, 20 ml lidocaine 1% and 4 mg dexamethasone; group C with 20 ml ropivacaine 0,5%, 20 ml lidocaine 1% and 8 mg dexamethasone.

All groups received postoperative analgesia when visual analog scale (VAS) over 3 (by request), with IV Perfalgan 1 g and morphine (loading dose 0.1 mg/kg and titration until VAS under 3, followed by subcutaneous (SC) administration of 1/2 of total loading dose on demand for the following 24 hours (h) .

Efficacy was evaluated by the time interval from performing the block until the first analgesic dose required, the total amount of morphine in the first 24 h postoperative, the patient satisfaction and the neurological side effects.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* BMI<40

Exclusion Criteria:

* High risk grade hypertension
* Chronic renal failure
* Known allergy to drugs used
* Chronic treatment with steroids
* Drugs dependency
* History of diabetes mellitus
* Ulcer or chronic gastritis
* Infection on the puncture site
* Neuropathy at the surgical level
* Coagulopathy
* Requesting another type of anesthesia
* Fear to sign informed consent
* By-pass aorto-femoral

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2015-11; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
the total amount of morphine | At 24 hour postoperative
  the morphine administered in milligrams

SECONDARY OUTCOMES:
the patient satisfaction | At 24 hour postoperative
  evaluation of satisfaction by a questionnaire
the number of patients with neurological motility side effects | At 24 h postoperative
  Following the postoperative motility of operated lower limb by Bromage scale
duration of analgesia | the first 24 hours
  the time interval from performing the block until the first analgesic dose required at VAS >3 (0 - no pain, 10 - the worst pain possible
the number of patients with neurological sensibility side effects | At 21 days postoperative
  Following postoperative sensibility of operated lower limb by pinprick test

CONTACTS AND LOCATIONS:
Overall Officials: Ioan Cristian Stoica, Prof, Study Director — Foisor Orthopedics Clinical Hospital
Locations (1):
- Foisor Orthopedics Clinical Hospital, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huynh TM, Marret E, Bonnet F. Combination of dexamethasone and local anaesthetic solution in peripheral nerve blocks: A meta-analysis of randomised controlled trials. Eur J Anaesthesiol. 2015 Nov;32(11):751-8. doi: 10.1097/EJA.0000000000000248. PMID 25774458
- [Result] Williams BA, Hough KA, Tsui BY, Ibinson JW, Gold MS, Gebhart GF. Neurotoxicity of adjuvants used in perineural anesthesia and analgesia in comparison with ropivacaine. Reg Anesth Pain Med. 2011 May-Jun;36(3):225-30. doi: 10.1097/AAP.0b013e3182176f70. PMID 21519308
- [Result] De Oliveira GS Jr, Castro Alves LJ, Nader A, Kendall MC, Rahangdale R, McCarthy RJ. Perineural dexamethasone to improve postoperative analgesia with peripheral nerve blocks: a meta-analysis of randomized controlled trials. Pain Res Treat. 2014;2014:179029. doi: 10.1155/2014/179029. Epub 2014 Nov 18. PMID 25485150
- [Result] Brummett CM, Williams BA. Additives to local anesthetics for peripheral nerve blockade. Int Anesthesiol Clin. 2011 Fall;49(4):104-16. doi: 10.1097/AIA.0b013e31820e4a49. PMID 21956081
- [Result] Williams BA, Schott NJ, Mangione MP, Ibinson JW. Perineural dexamethasone and multimodal perineural analgesia: how much is too much? Anesth Analg. 2014 May;118(5):912-4. doi: 10.1213/ANE.0000000000000203. No abstract available. PMID 24781562